CLINICAL TRIAL: NCT05010018
Title: A Mobile Application to Improve Procurement and Distribution of Healthful Foods & Beverages in Low Income Urban Communities
Brief Title: A Mobile Application to Improve Procurement and Distribution of Healthful Foods & Beverages in Baltimore City
Acronym: BUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R34HL145368 (NIH); R34HL145368 (NIH)
Record Dates: First submitted 2021-07-22; First posted 2021-08-18 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): We will pilot the BUD app in 19 intervention corner stores over an 8-month period in East Baltimore. During this time, we will collect data from corner store owners, producers, whole salers, and consumers.
  Interventions: Behavioral: Web-based application connecting small food store owners and suppliers of healthier foods and beverages
- Control (No Intervention): We will collect data from 19 control corner stores over the same 8-month period. They will not receive any form of intervention or delay intervention.

INTERVENTIONS:
Behavioral: Web-based application connecting small food store owners and suppliers of healthier foods and beverages — The primary intervention is a web-based app that connects small food store owners in low income Baltimore with suppliers of healthier foods and beverages. To reduce costs associated with small purchasing quantities by corner stores, and high delivery charges, the BUD app uses collective purchasing and shared delivery strategies. BUD will be implemented in four stages, where each stage promotes different food/beverage items and introduces new features. The app will be bundled with a small subsidy in stages 1-2 to encourage initial use, increase familiarity with the app and reduce risk. Trainings in the use of the app will take place at the beginning of each phase. BUD will use collective purchasing at stage 2 of implementation (BuddyUp!). The BuddyLift! feature will start in stage 3, enabling small store owners to deliver BuddyUp! deals to other stores for an additional discount. Participating stores and wholesalers will receive point of purchase materials to promote BUD products.
  Arms: Intervention

SUMMARY:
Low-income urban communities have many small food stores, but poor access to healthier foods and beverages. The investigators will develop, implement and evaluate the feasibility of a Baltimore Urban food Distribution (BUD) web-based application (app) to improve access to affordable, healthier products from local producers/wholesalers in 38 urban corner stores in low-income Baltimore neighborhoods, using a randomized controlled trial design and assess its impact on store stocking and sales. The R34 will provide a developed and tested version of the BUD app, which will resolve challenges related to affordability and delivery of healthful foods and beverages to small food stores, permit development of new instruments, assess potential impacts at the consumer level, permitting power and sample size estimates for the full-scale clinical trial, and demonstrate the investigators' ability to recruit and retain large numbers of wholesalers, producers, and corner stores in low-income urban settings.

DETAILED DESCRIPTION:
The overarching goal of this application is to develop and pilot test a web-based application (app) that will increase access to healthier foods and beverages in low-income urban communities in the United States. Small retail food stores are ubiquitous in low-income urban settings throughout the US and present a unique opportunity to supply surrounding neighborhoods with healthful food options. However, these small stores usually carry few or no foods that are both healthy and affordable. A primary barrier to stocking healthy, affordable foods in small urban food stores is the lack of an adequate distribution network; small store owners generally need to travel on their own to obtain healthy foods and beverages for their stores. Low access to healthy food and high access to food with low nutritional value have been associated with poor diet quality, obesity and chronic disease in many studies.

The study team has worked for more than 17 years in Baltimore to develop, implement, and evaluate chronic disease prevention programs by improving the food environment in low-income communities. The investigators' preliminary formative research assessed the initial acceptability of a mobile app that will enable small urban food store owners to access a range of healthy foods from local wholesalers and producers, and facilitate affordable delivery to their stores. The study team found high acceptability for an app that would leverage the collective purchasing power of digitally-networked small food stores and introduce cost efficiencies into food delivery. For this NHLBI Clinical Trial Pilot Study (R34), the investigators propose to develop a working web-based Baltimore Urban food Distribution (BUD) app, pilot the app, and evaluate its feasibility and impact on the availability, prices and distribution of healthful foods and beverages in East Baltimore, with the following primary aims: 1) To develop and optimize a technically stable and functional digital strategy to overcome small retail food system constraints common in low-income urban food settings; 2) To pilot the BUD app with Baltimore-based producers/wholesalers and corner stores, and assess its feasibility (i.e., acceptability, operability, perceived sustainability, user satisfaction); and 3) To evaluate the impact of the BUD app on corner store stocking (availability, timeliness, quality), prices, and sales of healthy and unhealthy foods and beverages in a pilot study employing a randomized controlled trial design of 38 corner stores. Secondary aims will examine impact on consumers and a cost-benefit analysis for participating retailers and producers.

Findings will permit the investigators to: 1) produce a functional and acceptable web-based app, 2) provide preliminary data needed for power calculations for the full-scale trial, 3) generate and refine process evaluation instruments and set standards for implementation, and 4) establish protocols and demonstrate the study team's ability to recruit and retain large numbers of wholesalers, producers, corner stores and consumers. The study team will assess generalizability of the app by conducting feasibility assessments of the developed app with small store owners and suppliers in other urban settings. The findings from this R34 application are essential to support a full-scale clinical trial, which will test a multi-city deployment of the BUD app and assess its impact on obesity and diet.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for stores:

Store owner/manager willing and able to order food through a smart phone or other internet-enabled device

Store owner/manager willing to attend in-store trainings in the use of the BUD App

Store located in a low-income neighborhood considered as a Healthy Food Priority Area by the Johns Hopkins Center for a Livable Future111 in East Baltimore

Store located >0.25 miles from a supermarket

Store classified as a small food store (< 4 aisles, < 2 cash registers)

Store owner/manager is English, Korean, Spanish or Mandarin-speaking for first language

Inclusion criteria for wholesalers and producers:

Provide service to Baltimore City (e.g., for producers, this could mean participating in Baltimore City-based farmers markets)

Willing to use the BUD app, including posting and maintaining data on a minimum number of products

Willing to participate with delivery services arranged

Inclusion criteria for consumers (community members):

* Regular customers of the store (purchase food items at least once a week in the store) identified by the small food store owner/manager enrolled in the study
* Adult (between 21 years old and 75 years old)
* Live/work within a 1/2 mile radius from one of the 38 small food stores participating in the study
* Live in a household of at least 2 persons (criteria intended to provide a more stable sample, to reduce loss to follow-up)

Exclusion Criteria:

* Anticipate moving out of Baltimore City in the next 12 months
* Pregnant (due to changes in diet, weight and body composition)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Gittlesohn, PhD, Principal Investigator — Johns HopkinsUniversity
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests would be reviewed by the project steering committee (composed of study investigators and the appropriate NIH project officer). They will receive de-identified data spreadsheets with codebooks that explain the meaning of each variable and the corresponding codes for each variable. In addition, they will receive a detailed description of the study design.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: People may request data for research purposes, after data have been collected, cleaned, analyzed and the primary study outcome papers have been published.
Access Criteria: External parties would be required to complete an online request form, describing the specific datasets required, intended use/analyses, commitment to confidentiality, etc.

REFERENCES:
- [Derived] Lewis EC, Zhu S, Oladimeji AT, Igusa T, Martin NM, Poirier L, Trujillo AJ, Reznar MM, Gittelsohn J. Design of an innovative digital application to facilitate access to healthy foods in low-income urban settings. Mhealth. 2023 Nov 3;10:2. doi: 10.21037/mhealth-23-30. eCollection 2024. PMID 38323147
- [Derived] Gittelsohn J, Lewis EC, Martin NM, Zhu S, Poirier L, Van Dongen EJI, Ross A, Sundermeir SM, Labrique AB, Reznar MM, Igusa T, Trujillo AJ. The Baltimore Urban Food Distribution (BUD) App: Study Protocol to Assess the Feasibility of a Food Systems Intervention. Int J Environ Res Public Health. 2022 Jul 26;19(15):9138. doi: 10.3390/ijerph19159138. PMID 35897500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in 2021-2023 for corner stores and food-store consumers. Corner store recruitment occurred at the individual stores. Food-store consumer recruitment occurred via flyers at stores and on social media.
Pre-assignment Details: Of the 290 participants enrolled, 163 participants recruited into the study were later found out to be "bots" and thus their data was removed from the study and they were not assigned into study arms. 127 food-store consumers were assigned to the study arms. 20 stores were recruited into the study and 16 finished. 2 stores closed and 2 were converted into restaurants.
Units Other Than Participants: Corner stores
Groups:
- Intervention: Intervention corner-store; Consumers living within 3/4 of a mile of intervention store
- Control: Corner stores in the control arm do not receive the application. Consumers living more than 3/4 of a mile from intervention stores.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 16; 4 Corner stores | 111; 16 Corner stores
Corner-store Owners | 4; 4 Corner stores | 16; 16 Corner stores
Completed | 6; 2 Corner stores | 52; 14 Corner stores
Not Completed | 10; 2 Corner stores | 59; 2 Corner stores

BASELINE CHARACTERISTICS:
Population: Baseline demographic data were collected only for food-store consumer participants (n=290). No baseline or demographic data were collected for corner store owners or stores.
  Therefore, baseline characteristics are reported only for the consumer arms ("Intervention-Consumer" and "Control-Consumer"). The corner store owner arms ("Intervention: Corner store Owners" and "Control: Corner store Owners") are not included because no owner-level demographic data were collected.
Groups:
- Intervention- Consumer: Consumers living within 3/4 of a mile of intervention store
- Control-Consumer: Consumers living more than 3/4 of a mile from intervention stores.
- Total: Total of all reporting groups
Arm/Group | Intervention- Consumer | Control-Consumer | Total
Number analyzed (Participants) | 16 | 111 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 110 | 126
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 72 | 85
  Male | 3 | 39 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 10 | 55 | 65
  White | 5 | 44 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 11 | 11
  Not Hispanic or Latino | 14 | 85 | 99
  Unknown or Not Reported | 2 | 15 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Stocking of Healthy Foods as Assessed by a Store Impact Questionnaire
Description: Stocking of healthy foods will be assessed from Pre to Post intervention at participating corner stores. A Store Impact Questionnaire will capture the number of promoted foods and beverages stocked during each visit, based on direct structured observation of corner store shelves. The investigators will create healthy food availability scores (range 0-27). The investigators will calculate change scores, by subtracting each pre measure from each post measure. A higher score is better, indicates more healthy options became available over the intervention.
Time Frame: Up to 2 months prior to intervention; up to 2 months post intervention
Population: Corner-stores are the analysis group. Food-store consumers (participants) were not the analysis group for this outcome. The Overall Number of Participants Analyzed represents the number of corner-store owners for each Arm/Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Corner store
Groups:
- Control Cornerstore: Corner store that did not use the app
- Intervention Cornerstore: Cornerstore that used the app
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 14 | 2
Number analyzed (Corner store) | 14 | 2
score on a scale | -9.5 (3.5) | -2.2 (2.7)
Statistical Analysis 1: Comparison: Control Cornerstore vs Intervention Cornerstore; Test type: Other; p = 0.22, welch's t-test

2. Primary Outcome: Change in Sale of Healthy Foods
Description: Change in sale of promoted healthy foods will be assessed from Pre to Post intervention at participating corner stores (recall over the last 30 day period). Store owners will be asked to recall the sale of selected healthy foods over the last 30 day period.
Time Frame: Up to 2 months prior to intervention, up to 2 months post intervention
Population: Analysis population represents corner stores with both baseline and post-intervention data collected
Measure: Mean (Standard Deviation); unit: healthy foods
Units Other Than Participants: Corner store
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 5 | 1
Number analyzed (Corner store) | 5 | 1
healthy foods | -0.03 (0.58) | 0.50 (NA) — Standard deviation is NA because the intervention arm contains only one store owner

3. Secondary Outcome: Change in Purchasing of Healthy Foods by Consumers
Description: Adult consumer purchasing of healthy promoted foods and beverages will be captured by the adult impact questionnaire (AIQ) which will be conducted at baseline and post-treatment in a sample of 190 regular customers (5 customers/store in 19 intervention and 19 control stores). Customers will be requested to report how often they purchased specific healthy promoted foods and beverages in the past 7 days, and where these foods were purchased. A score called the "Healthy Food Purchasing Score" will be calculated and have a possible score value ranging from 0-38 points. We will subtract the pre score from the baseline score to calculate change in purchasing of healthy foods by consumers.
Time Frame: The Pre measure will be made in the two months prior to starting the intervention; the Post measure will be made in the two month after the end of the intervention
Reporting Status: Not Posted, anticipated posting 2026-04

4. Secondary Outcome: Change in Consumption of Healthy Eating Index by Consumers
Description: Adult customer consumption of healthy and unhealthy foods is captured by the semi-quantitative Block Food Frequency Questionnaire (FFQ) for the entire consumer sample. This validated questionnaire contains questions regarding the frequency and amount of consumption of over 50 commonly consumed foods. The Block FFQ has been validated for use in low income African American urban populations. Investigators will calculate a Healthy Eating Index (scoring ranging from 0-100) using the consumed food frequencies and portion sizes reported on the FFQ. The investigators will assess change in the consumption of healthy foods by subtracting the pre HEI score from the post HEI score.
Time Frame: The Pre-measure will be made in the two months prior to starting the intervention; the Post-measure will be made in the two month after the end of the intervention
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: Estimated Changes (Reduction) in Operating Costs
Description: Data collection will include a Supplier Fixed and Variable Costs spreadsheet completed by the store owners which will provide information for the cost-benefit analysis of the treatment for each sector of the Baltimore food system participating in the BUD study. Respondents will be asked to estimate changes in these operating costs from before use of the app to the present. The team will compute savings in operating costs and the unit of measurement will be U.S $. It will consider the fixed and variable costs. Fixed costs will include item costs that will not change with the level of activity (rent of space; interest in long-term loans;). Variable costs will include item costs that change with level of activity (labor expenses; material expenses, transportation costs, utilities).
Time Frame: Up to 2 months post intervention
Population: Analysis population represents corner stores with both baseline and post-intervention data collected
Measure: Mean (Standard Deviation); unit: US dollars
Units Other Than Participants: Corner store
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 5 | 1
Number analyzed (Corner store) | 5 | 1
US dollars | 4.00 (0.71) | 3.00 (NA) — Standard deviation is NA because the intervention arm contains only one store.

6. Secondary Outcome: Estimated Changes (Savings) in Acquisition Prices
Description: The Supplier Fixed and Variable Costs spreadsheet completed by the store owners will provide information for the cost-benefit analysis of using the BUD app for each participating sector of the Baltimore food system. The quantity and price of acquisition will be observed and used to compute the total savings. The unit of measurement will be US dollars.
Time Frame: Up to 2 months post intervention
Population: Analysis population represents corner stores with both baseline and post-intervention data collected
Measure: Mean (Standard Deviation); unit: US dollars
Units Other Than Participants: Corner store
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 5 | 1
Number analyzed (Corner store) | 5 | 1
US dollars | 3.8 (0.84) | 5.0 (NA) — Standard deviation is NA because the intervention arm contains only one store.

7. Secondary Outcome: Estimated Total Financial Expenses
Description: The Supplier Fixed and Variable Costs spreadsheet completed by the store owners using the BUD app will provide information for estimated changes in total financial expenses. This data collection will include the financial costs of acquiring and implementing the BUD application. It will consider the fixed and variable costs. Fixed costs will include item costs that will not change with the level of activity (rent of space; cost items that need to be paid even if the producer close). Variable costs will include item costs that change with level of activity (labor expenses; material expenses, transportation costs, utilities). The unit of measurement will be U.S $ monthly, with adjustment (e.g., by total products).
Time Frame: Up to 2 months post intervention
Population: Analysis population represents corner stores with both baseline and post-intervention data collected
Measure: Mean (Standard Deviation); unit: US dollars
Units Other Than Participants: Corner store
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 5 | 1
Number analyzed (Corner store) | 5 | 1
US dollars | 3.6 (0.55) | 5.0 (NA) — Standard deviation is NA because the intervention arm contains only one store.

8. Secondary Outcome: Changes in Prices of Healthy Foods
Description: Prices of healthy promoted foods and beverages will be collected 5x, as well as of a subset of less healthy alternatives. The SIQ and process evaluation instruments will capture the price of each product during each visit, based on corner store owner report. Most corner stores do not label individual foods with the price, nor are shelves labeled. The investigators have successfully collected pricing information using this method for previous studies in Baltimore corner stores. The investigators will examine changes in prices from the point the food is sold at the store, until the end of the intervention. A change score will be calculated by subtracting the pre price from the post price of each healthy food. The investigators will use this information to compare prices of these healthier foods with those of unhealthy alternatives to help ensure acceptability to customers.
Time Frame: Up to 2 months prior to intervention, up to 2 months post intervention
Population: Analysis population represents corner stores with both baseline and post-intervention data collected
Measure: Mean (Standard Deviation); unit: US dollars
Units Other Than Participants: Corner store
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 5 | 1
Number analyzed (Corner store) | 5 | 1
US dollars | 3.6 (0.89) | 2.0 (NA) — Standard deviation is NA because the intervention arm contains only one store

9. Secondary Outcome: Change in Feasibility Metrics: App Satisfaction, Acceptability, Operability, and Perceived Sustainability as Assessed by Survey
Description: Store-owner satisfaction with the BUD app was collected at two time points: pre-intervention (baseline) and post-intervention. Corner store owners using the BUD app were asked to rate their agreement with multiple statements related to app usability, perceived benefit, operational feasibility, and competitive advantage. Each item used a 5-point Likert response scale (1 = strongly disagree to 5 = strongly agree), the total composite score ranges from 3-15 with higher scores better, indicating greater satisfaction. A composite satisfaction score was calculated at each time point, and change was computed as the post-intervention score minus the baseline score.
Time Frame: Pre-intervention (baseline) up to approximately one year following completion of the intervention.
Population: Analysis population represents corner store owners with both baseline and post-intervention data collected
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Cornerstore | Intervention Cornerstore
Number analyzed (Participants) | 5 | 1
Score on a scale | -0.133 (1.17) | 1.667 (NA) — Standard deviation is NA because the intervention arm contains only one store owner

10. Secondary Outcome: Process Metrics: Reach as Assessed by Intervention Corner-store Owners Who Participate in the Trial
Description: During intervention delivery, the investigators will assess multiple process evaluation metrics. These will be recorded via in-person data collection, or through the BUD app itself. The first process measures is reach which is measured by the # intervention store owners who actively participate in trial ( # who access BUD app at least once).
Time Frame: Pre-intervention (baseline) up to 1 year following completion of the intervention.
Population: Corner-store owners with data collected in the intervention arm who received and used the app
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Cornerstores that received the BUD App
- Control: Corner stores that did not use the BUD application
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 0
Participants | 4 | 0

11. Secondary Outcome: Process Metrics: Dose Delivered
Description: During intervention delivery, the investigators will assess multiple process evaluation metrics. These will be recorded via in-person data collection, or through the BUD app itself. The second process measure is dose delivered which includes # trainings completed by JHU team/# planned, # promotional materials posted/# planned, and # subsidies provided/# planned.
Time Frame: Measures collected during the trial will occur at pre-intervention, during the intervention and immediately after the intervention
Reporting Status: Not Posted, anticipated posting 2026-04

12. Secondary Outcome: Process Metrics: Fidelity
Description: During intervention delivery, the investigators will assess multiple process evaluation metrics. These will be recorded via in-person data collection, or through the BUD app itself. The third process measure is fidelity which includes such measurements as # store owners actively using the BUD app, # times they use the app, and # using materials/subsidies provided.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 2 years
Description: Consumers and Store-owners were followed for adverse events
Groups:
- Intervention: Corner store owners using the application, Consumers living within 3/4 of a mile of intervention store
- Control: Corner store owners not using the application, Consumers living more than 3/4 of a mile from intervention stores.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/127
Other Adverse Events (participants affected / at risk) | 0/20 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Stat Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT05010018/Prot_SAP_000.pdf